CLINICAL TRIAL: NCT04890522
Title: A Randomized, Open-label, Multicentre, Phase II/III Study of Low-dose Long-term Continuous Intravenous Infused 5-fluorouracil Versus Gemcitabine Combined With Cisplatin and JS001 as First-line Therapy for Metastatic Nasopharyngeal Carcinoma
Brief Title: An Open-label, Multicentre, Phase II/III RCT of PFLL Versus GP Combined With JS001 as the First-line Therapy for mNPC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-409-01
Record Dates: First submitted 2021-05-04; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Nasopharyngeal Carcinoma; Metastasis; Chemotherapy; Immunotherapy; Survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Cisplatin; Fluorouracil; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 5-fluorouracil intravenous infusion at 200mg/m2/d for 30 continuous days, and intravenous infusion of cisplatin 80 mg/m2 on day 1 and day 28, and intravenous infusion of JS001 240mg on day 1 and day 21, every 60 days.
  Interventions: Drug: Triprilimab(JS001); Drug: Cisplatin; Drug: 5-Fluorouracil
- Control group (Active Comparator): gemcitabine at a dose of 1,000 mg/m2 by intravenous infusion on days 1, 8, and intravenous infusion of cisplatin at a dose of 80 mg/m2 on day 1, and intravenous infusion of JS001 240mg on day 1, every 21 days.
  Interventions: Drug: Triprilimab(JS001); Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Triprilimab(JS001) — Maximum 6 cycles for combined therapy and maintenance for up to 2 years.
Drug: Cisplatin — Maximum 6 cycles for combined therapy.
Drug: 5-Fluorouracil — Maximum 6 cycles for combined therapy.
  Arms: Experimental group
Drug: Gemcitabine — Maximum 6 cycles for combined therapy.
  Arms: Control group

SUMMARY:
The treatment of distant metastasis is a key challenge for nasopharyngeal carcinoma because of poor outcomes, among which, chemotherapy is the cornerstone. However, many studies reported the use of different chemotherapy regimens to prolong the survival of metastatic nasopharyngeal carcinoma, while few of them focused on how to reduce the side effects of chemotherapy or improve the life quality of patients. Blocking the immune checkpoint is one of the effective strategies of tumor immunotherapy. Thus, we sought to find a proper chemotherapy regimen combined with PD-1 antibody JS001.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal carcinoma diagnosed by pathology or cytology.
* Primarily metastatic (stage IVB as defined by the International Union against Cancer and American Joint Committee on Cancer staging system for NPC, eighth edition) is not amenable for local-regional treatment or curative treatment.
* Has not received prior systemic treatment for metastatic nasopharyngeal carcinoma, except for neoadjuvant chemotherapy, concurrent chemoradiotherapy, or adjuvant chemotherapy 6 months prior to the first treatment.
* The Karnofsky performance status score is at least 70 points (if the decreased score is caused by the tumor, the minimum score can be 50 points after the judgment of researchers.)
* Has at least one measurable target lesion based on RECIST v1.1, which is never received local treatment like radiotherapy.
* Life expectancy ≥ 3 months.
* The lab examination results of the screening must fulfill all of the following (use of any blood components, hematopoietic stimulating factors, etc. are not allowed within 14 days before screening):

  1. absolute neutrophil count ≥1.5×10^9/ L;
  2. platelet count ≥ 100×10^9/ L;
  3. hemoglobin ≥ 8.0 g/dL;
  4. serum albumin ≥ 2.8g/dL;
  5. aspartate transferase(AST) and alanine transferase(ALT) ≤ 1.5 ×ULN; total bilirubin ≤ 1.5×ULN (if has liver metastasis, AST and ALT ≤ 5×ULN);
  6. creatinine clearance >50 mL/min.
* Men with reproductive capacity or women of childbearing potential must use highly effective contraceptive methods during the trial (e.g., oral contraceptives, intrauterine device, sexual abstinence or barrier method combined with spermicide), and continue contraception for 3 months after the last injection of JS001 and 6 months after the end of chemotherapy.
* Has signed the Informed Consent Form.

Exclusion Criteria:

* Allergic to monoclonal antibodies, any JS001 components, gemcitabine, cisplatin, or 5-fluorouracil.
* Has prior therapy including anti-PD-1, anti-PD-L1, or CTLA4.
* Major surgery within 28 days prior to the randomization (not including diagnostic surgery) or plan to be conducted during the study.
* Active autoimmune disease requiring systemic treatment or has a history of autoimmune disease.
* Requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment.
* Allergic to macromolecular protein preparation ingredients.
* Has central nervous system (CNS) metastasis with clinical symptoms.
* Had other invasive malignant diseases, except excised basal-cell skin carcinoma, cervical carcinoma in situ, or other cancers curatively treated more than 5 years before study entry.
* Has cardiac clinical symptoms or disease out of control.
* Has an active infection or unexplained fever with more than 38.5 ℃ during screening and prior to first administration.
* Has acquired or congenital immune-deficient disease, or active hepatitis.
* History of drug abuse or alcohol abuse.
* The investigator judges other factors that may lead to the forced termination of this study, including but not limited to: other serious conditions (including mental disorder) that require concomitant treatment, severe laboratory test abnormalities, family or social factors that may affect the safety of patients or the collection of trial data and samples.
* Pregnancy or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 622 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 5 years
  Progression-free survival
OS | Up to 5 years
  Overall survival
Severe drug-related adverse events | Up to 2 approximately years
  grade III-V according to CTCAE v4.0

SECONDARY OUTCOMES:
ORR | Up to 2 approximately years
  Objective response rate
DCR | Up to 2 approximately years
  Disease control rate
DOR | Up to 2 approximately years
  Duration of response
Minor drug-related adverse events | Up to 2 approximately years
  grade I-II according to CTCAE v4.0
Quality-adjusted survival | Up to 5 years
  Quality-adjusted Time Without Symptoms of disease or Toxicity of treatment (Q-TWiST), a measure involving the partitioning of survival duration into clinically relevant health states (e.g., treatment toxicity, disease progression, progression-free), assigning preference weights (or utilities) to these health states, and calculating quality of life-adjusted weighted sums of the mean duration of each health state to create the overall Q-TWiST scores.
Therapeutic gain | Up to 2 approximately years
  Calculated by dividing person-year rate of overall survival by person-year rate of serious toxicity.
Incremental Cost-Effectiveness Ratio (ICER) | Up to 2 approximately years
  To estimate the costs and health gains of different interventions, calculated as incremental cost divided by life years gained.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No